CLINICAL TRIAL: NCT00075439
Title: A Phase II Trial of ZD1839 (Iressa®) in Metastatic Neuroendocrine Tumors
Brief Title: Gefitinib in Treating Patients With Progressive Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02796; MC0279; N01CM62205 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Metastatic Gastrointestinal Carcinoid Tumor; Pancreatic Polypeptide Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Somatostatinoma; WDHA Syndrome
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Carcinoma, Islet Cell; Somatostatinoma; Vipoma | interventions — Gefitinib

ARMS (1):
- Arm I (Experimental): Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well gefitinib works in treating patients with progressive metastatic neuroendocrine tumors. Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 6 month progression free survival rate in patients with progressive, advanced neuroendocrine tumors treated with ZD1839.

SECONDARY OBJECTIVES:

I. Objective tumor response rate. II. Progression free survival and time to progression. III. Improvement in circulating hormone levels. IV. Overall survival V. We will explore the molecular characterization of these tumors in attempt to understand the role of EGFR expression and its inhibition with ZD1839 in neuroendocrine tumors. The measurements will be performed on pretreatment and post-treatment tumor biopsies when possible: EGFR expression and gene amplification (IHC for EGFR and phosphorylated EGFR, ISH for gene amplification); Activation of the Ras/Raf/MAPK pathway (IHC for phosphorylated MAPK); Cell proliferation (Ki-67 staining); Apoptosis (TUNEL assay).

OUTLINE: This is a multicenter study. Patients are stratified according to disease type (carcinoid vs islet cell and other neuroendocrine tumors).

Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 2 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic neuroendocrine neoplasms or histologic confirmation of primary neuroendocrine tumor with clear clinical evidence of metastases
* Measurable disease
* Radiographic evidence of disease progression, following any prior systemic therapy, chemoembolization, embolization, or observation; for eligibility purposes, disease progression will be defined as follows:

  * Either of the following documented by comparison of the on-study radiographic assessment with a prior assessment of the same type performed within the previous 60 calendar weeks:

    * Appearance of a new lesion
    * At least 20% increase in the longest diameter (LD) of any previously documented lesion or an increase in the sum of the LDs of multiple lesions in aggregate of 20%
* ≥4 weeks from the completion of major surgery, chemotherapy or other systemic therapy and hepatic artery embolization/chemoembolization to study registration
* ≥3 weeks from the completion of radiation therapy to study registration
* Recovered sufficiently from side effects of prior therapy
* Absolute neutrophil count (ANC) ≥ 1000/mm3
* PLT ≥ 75,000/ mm3
* Hgb ≥ 8.0 g/dL
* Total bilirubin ≤ 2 x upper normal limit (UNL)
* Alkaline phosphatase ≤ 3 x UNL (5 x UNL if liver metastases present)
* AST ≤ 3 x UNL (≤ 5 x UNL if liver metastases present)
* Creatinine ≤ 1.5 x UNL
* ECOG performance score (ps) ≤ 2
* Life expectancy ≥ 24 weeks
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent

Exclusion Criteria:

* Thyroid carcinoma of any histology or pheochromocytoma/paraganglioma
* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
  * NOTE: The effects of the agent(s) on the developing human fetus at the recommended therapeutic dose are unknown
* Anaplastic or high-grade histology
* Any of the following prior therapies:

  * > 1 prior systemic chemotherapy regimen (chemoembolization not counted as systemic chemotherapy)
  * Prior EGFR targeted regimen (e.g. OSI-774, EKB-569, ZD1839)
  * < 4 weeks from last Interferon injection
  * < 2 weeks from last octreatide short acting injection or < 6 weeks long acting injection; Note: concurrent octreatide allowed if stable dose has been administered for ≥1 month, there is documented tumor progression on the current dose, and there is no current plan for increasing dose • Other concurrent treatment considered investigational
* Concurrent chemotherapy or radiation therapy
* Any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication (e.g. dysphagia or inability to swallow capsules intact).
  * Requirement for IV alimentation
  * Prior procedures clearly adversely affecting intestinal absorption
  * Active peptic ulcer disease
  * Failure to fully recover from adverse effects of prior therapies regardless of interval since last treatment
* Known abnormality of cornea, such as:

  * History of dry eye syndrome or Sjogren syndrome
  * Congenital abnormality
  * Abnormal slit-lamp examination using a vital dye (e.g.: fluorescein or Bengal-rose)
  * Abnormal corneal sensitivity test (Schirmer test)
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptoms of congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirement
* Known brain metastases; Note: These patients are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Known HIV-positive patients receiving combination anti-retroviral therapy; Note: These patients are excluded from the study because of possible pharmacokinetic interactions with ZD1839 and because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination and anti-retroviral therapy when indicated
* Concurrent or recent use (≤ 7 days prior to ZD1839 administration) of phenytoin, carbamazepine, barbiturates, rifampicin, oxcarbazepine, rifapentine, modafinil, or St. John's Wort; Note: Because these drugs induce CYP3A4 enzymes and can cause reductions in ZD1839 plasma concentrations below levels thought to be biologically active, patients with concurrent or recent use of these drugs are excluded from the study
* History of other invasive malignancy ≤ the previous 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2003-12; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients progression-free at 6 months | At 6 months
  If patients are lost to follow-up or discontinue active monitoring prior to 6 months post-registration, we will consider censoring them for the evaluation of the primary endpoint. Here, Kaplan-Meier methodology will be used to estimate the final success proportion (ie, 6 month success rate with a 95% confidence interval). Otherwise, ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Incidence of adverse events graded according to NCI CTCAE version 3.0 | Up to 2 years
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Confirmed tumor response to treatment will be evaluated and will be considered a PR or CR on consecutive evaluations at least 4 weeks apart | Up to 2 years
  The proportion of responses will be evaluated and will be tabulated. Assuming a binomial distribution for the incidence of response, 95% confidence intervals will also be generated.
Survival time | Time from registration to death due to any cause, assessed up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from randomization to documentation of disease progression, assessed up to 2 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of response | Date from which the patient's objective status is first noted to be either a CR or PR to the date progression is documented, assessed up to 2 years
  This data will be descriptively summarized and graphically evaluated.
Time to treatment failure | Time from the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, refusal, or death, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Hobday, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States